CLINICAL TRIAL: NCT03178760
Title: Determination of Normal Measures of Optic Nerve Sheath Diameter in Children
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ozlem Tolu Kendir, Fellow, Cukurova University
Other Study IDs: AU-70904504/393-19.06.2020
Record Dates: First submitted 2017-06-04; First posted 2017-06-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Optic Papilla Edema
Keywords: Optic nerve sheath diameter; average optic nerve sheath diameter for healthy children
MeSH Terms: conditions — Papilledema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonic Measurement will be taken from optic nerve sheat diameter and compared-classified. — Ultrasonic Measurement will be taken from optic nerve sheat diameter and compared-classified. Classifications will be done for;
  1. Age
  2. Gender
  3. Weight
  4. Length
  5. Waist Circumference
  6. Body mass index

SUMMARY:
The purpose of this study is to measurement of optic nerve sheath diameter in children without intracranial pressure increase and determine the average optic nerve sheath diameters for healthy children.

DETAILED DESCRIPTION:
The purpose of this study is to measurement of optic nerve sheath diameter in children without intracranial pressure increase and determine the average optic nerve sheath diameters for healthy children. For that, between 4 and 18 years old children will be selected. After taking of measurements, following parameters will be taken into account and measurements will be classified with those parameters .

1. Age
2. Gender
3. Length (cm)
4. Weight (kg)
5. Waist Circumference (cm)
6. Body Mass Index

ELIGIBILITY:
Inclusion Criteria:

• Children without cerebral edema.

Exclusion Criteria:

• Children with cerebral edema.

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Gender Based: Yes — Measurements will be classified with gender.
Study Population: all patients without cerebral edema applied the emergency care unit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Measurement of optic nerve sheath diameter | 1-3 minute
  mm

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided